CLINICAL TRIAL: NCT02385994
Title: A Prospective Multi-Center Study of a Novel Dual-Wavelength, Dual-Pulse Duration Laser for the Treatment of Melasma and Lentigines in Asian Skin
Brief Title: A Prospective Multi-Center Study Using Laser for the Treatment of Melasma and Lentigines in Asian Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-14-EN01
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Melasma; Lentigines
MeSH Terms: conditions — Melanosis; Lentigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- enLighten Laser Treatment (Experimental): Melasma, Cohort I or Lentigines, Cohort II will be treated with dual-pulse duration, dual-wavelength 532nm KTP/1064nm Nd:YAG laser.
  Interventions: Device: enLighten Laser
- Control (No Intervention): Melasma subjects randomized to non-treatment will receive no treatments.

INTERVENTIONS:
Device: enLighten Laser — enLighten Laser treatment with dual-pulse width and dual-wavelength
  Arms: enLighten Laser Treatment

SUMMARY:
The purpose of this investigation is to evaluate safety and efficacy of the Cutera enlighten dual-pulse duration, dual-wavelength 532nm KTP/1064nm Nd:YAG laser for the treatment of melasma and lentigines on the face in Asian skin.

DETAILED DESCRIPTION:
This is a multi-center prospective, 2 cohort study in 80 male or female subjects of Asian-descent, who desire laser treatment for moderate to severe melasma (all types) or lentigines (all types) located on the face. Forty subjects will be enrolled in cohort 1 and randomized to either treatment or control arm. Forty subjects will be enrolled for treatment of facial lentigines in cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 20 to 75 years of age (inclusive).
* Fitzpatrick Skin Type III - V.
* Has moderate to severe melasma (any type), OR any type of lentigo/lentigines ≥ 6mm in diameter, and desires laser treatment.
* Willing to refrain from using topical and systemic corticosteroids or retinoids, and topical or systemic prescription skin-lightening medications, except permitted topical steroid use as directed by study doctor.
* Willing to maintain consistent skin care regimen on the treatment area for the duration of the study, including the follow-up period.
* Must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Willing to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treatment area every day for the duration of the study, including the follow-up period.
* Willing to have digital photographs taken of the treatment area.
* Agree not to undergo any other procedure(s) in the treatment area during the study.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

* Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
* Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as laser or light-based procedures or surgery.
* Prior injection of collagen, hyaluronic acid filler or any other dermal filler in the target area within 6 months of study participation.
* Has mild melasma OR facial lentigo/lentigines less than 6mm in diameter.
* History of refractory melasma.
* History of allergy to local anesthetics, as applicable.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of hormone treatment, such as estrogen, progesterone and/or oral contraceptives, initiated within 3 months of study participation, or planning to discontinue hormone therapy during the study, as applicable.
* Systemic use of any prescription skin-lightening agent (such as tranexamic acid), isotretinoin (or other retinoid), photo-sensitizing medication, or corticosteroid within 6 months of and during study participation, except if the subject undergoes a 6-month wash-out period of excluded systemic prescriptions prior to first laser treatment.
* Topical use of any prescription skin-lightening agent (such as hydroquinone), isotretinoin (or other retinoid), photo-sensitizing medication, or corticosteroid on the treatment area within 6 months of and during study participation, except permitted topical steroid use as directed by study doctor and if subject undergoes a 6-month wash-out period of excluded topical prescriptions prior to first laser treatment.
* Anytime in life, had used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Investigator Assessment measured by 5-point improvement scale | 12 weeks
  Degree of improvement in melasma or lentigines at 3 months post-final treatment measured by 5-point improvement scale.

SECONDARY OUTCOMES:
Subject Assessment measured by 5-point improvement scale | 12 weeks
  Degree of improvement in melasma or lentigines at 3 months post-final treatment measured by 5-point improvement scale.
Melasma Subject's MASI Improvement | 12 weeks
  Change in mean Melasma Area and Severity Index (MASI) value at 3 months post-final treatment as compared to baseline
Relative Melanin Index | 12 weeks
  Change in mean relative Melanin Index (MI) value at 3 months post-final treatment as compared to baseline as assessed by mexameter measurements
Pain and Adverse Events | Day 1
  Incidence and severity of adverse device effects during the study period, including subject pain level during laser treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hin-Lee Chan, M.D., Ph.D, Principal Investigator — Hong Kong Dermatology and Laser Centre; Kei Negishi, M.D., Ph.D, Principal Investigator — Tokyo Women's Medical University
Locations (2):
- Hong Kong Dermatology and Laser Centre, Hong Kong, China
- Aoyama Institute of Women's Medicine, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided